CLINICAL TRIAL: NCT00049140
Title: Pilot Study of the Relationship Between EF5 Uptake and Concentration of Oxygen-Related Metabolites in Head and Neck Cancer
Brief Title: EF5 Compared With Other Methods of Detecting Oxygen Levels in Tumor Cells of Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M. Brizel, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David M. Brizel, MD, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000257828; DUMC-3512-02-3; NCI-5929
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Flow Cytometry; Immunohistochemistry; Biopsy

ARMS (1):
- EF5 (Experimental): This is a non randomised single arm pilot study.
  Interventions: Drug: EF5; Other: bioluminescence; Other: flow cytometry; Other: immunohistochemistry staining method; Procedure: biopsy

INTERVENTIONS:
Drug: EF5
Other: bioluminescence
Other: flow cytometry
Other: immunohistochemistry staining method
Procedure: biopsy

SUMMARY:
RATIONALE: Diagnostic procedures using the drug EF5 to detect the presence of oxygen in tumor cells may help to plan effective treatment for solid tumors.

PURPOSE: Phase II trial to compare diagnostic procedures using EF5 to that of other methods of detecting oxygen levels in tumor cells of patients who have head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the distribution, degree, and intrapatient and interpatient heterogeneity of hypoxia, as measured by EF5 binding in tumor tissue, in patients with head and neck cancer.
* Determine the distribution and intrapatient and interpatient heterogeneity of CA9 expression, as measured immunohistochemically, in these patients.
* Determine the distribution, concentration, and intrapatient and interpatient heterogeneity of glucose and lactate, as measured by bioluminescence imaging, in these patients.
* Determine whether there is spatial coordination between concentrations of lactate and glucose and the location of tissue hypoxia in these patients.
* Determine whether there is spatial coordination between the location of CA9 with hypoxia and/or lactate concentrations in these patients.

OUTLINE: Patients receive EF5 IV over 1-2.5 hours on day 1. Within 24-55 hours after EF5 infusion, patients undergo surgery.

Tumor tissue samples are examined for EF5 binding by immunohistochemistry, bioluminescence imaging, and flow cytometry.

Patients are followed at 1 month and then for survival.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck
* Clinically detectable disease by physical examination or radiographic studies
* Scheduled to undergo surgical resection of tumor or radiotherapeutic treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL

Renal

* Creatinine no greater than 1.8 mg/dL

Other

* No allergy to IV contrast dye
* No prior grade III or IV peripheral neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 week after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Concurrent radiotherapy allowed

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-08; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Heterogeneity of hypoxia as measured by EF5 binding at completion of accrual | One Year
Heterogeneity of CA9 expression by immunohistochemistry at completion of accrual | One year
Heterogeneity of glucose and lactate by bioluminescence imaging at completion of accrual | One Year
Spatial coordination as measured by EF5 binding at completion of accrual | One Year
Compare spatial coordination between the location of CA9 and hypoxia and/or lactate concentration at completion of accrual | One year

CONTACTS AND LOCATIONS:
Overall Officials: David M. Brizel, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States